CLINICAL TRIAL: NCT07350265
Title: Prospective Study Evaluating the Effectiveness of Intraoperative Ventilation for Predicting Postoperative Air Leaks During Major Lung Resections by Conventional or Robotic Thoracoscopy
Acronym: NODRAIN
Status: Not yet recruiting | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: COS-RGDS-2024-06-015-P-GRIGORO
Record Dates: First submitted 2025-09-22; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Air Leak From Lung; Lung Surgery
Keywords: intraoperative ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No intervention : Observational Cohort

SUMMARY:
Air leak from lung after major pulmonary resections is alveolar-pleural microfistulas resulting from damage to the visceral pleura during lung surgery. Despite advances in stapling techniques and repair methods to ensure pulmonary tightness after excision, air leak is the most common cause of prolonged hospital stay after lung surgery, accounting for 20 to 30% of post-surgical adverse events.

Although painless, they remain a significant source of morbidity. 10 to 20% of patients may have a prolonged air leak requiring intervention. Prolonged air leak is defined as an air leakage that persists for 5 days or more. Prolonged air leak is independently associated with increased hospitalization costs of 18% to 27% according to the series reported in the literature, but also with increased costs after hospital discharge, up to 90 days postoperatively.

Traditionally, the detection of air leak at the end of surgery is done by testing the lung for submersion in saline solution. With the development of major pulmonary resection techniques by conventional or robotic thoracoscopy (with closed chest), this method has become ineffective because it requires re-ventilating the lung in a closed rib cage, which cancels the visibility of the camera. However, the frequency of these adverse events and the morbidity associated with them now induces the placement of post-operative drains, which are very painful, unlike the leak itself, which makes the pain even more complex to bear for patients.

Given the rapid transition to a minimally invasive surgical approach, having a method to detect and quantify intraoperative air leak on a closed chest is necessary in order to accelerate patients' postoperative recovery, reducing their postoperative pain while controlling the incidence of complications.

A recent study has shown that the risk of postoperative air leak is possible based exclusively on intraoperative ventilator measurements, but the data are still too scarce to rely on them extensively.

DETAILED DESCRIPTION:
In this NODRAIN study, we aim to evaluate the effectiveness of intraoperative ventilation for the detection of intraoperative air leak from lung. Therefore, the main objective of this study is to investigate the effectiveness of intraoperative ventilation for the prediction of postoperative air leak.

Each patient will receive intraoperative ventilation, conducted for the diagnosis of air leak in routine practice, as well as their routine post-operative care, which is the installation of drains. The demonstration of a correlation will make it possible to determine a threshold for identifying patients for whom drainage would not be necessary, thus reducing their post-operative pain, the duration and the cost of hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Patient with pulmonary lobectomy or Anatomical segmentectomy with closed chest (conventional or robotic thoracoscopy);
* Patient affiliated with a health insurance scheme.
* Person who has not objected to the collection of his/her data for the purpose of the study.

Exclusion Criteria:

* Patient undergoing any type of lung resection by thoracotomy;
* Patient with a history of thoracic surgery on the same side;
* Patient with pulmonary fibrosis;
* Patient from a vulnerable population as defined in Articles L.1121-5 to 8 of the French Public Health Code.
* Patient undergoing conversion to thoracotomy;
* Patient undergoing conversion from planned pulmonary lobectomy or anatomical segmentectomy to atypical resection, bilobectomy or pneumonectomy;
* Drainage via two chest drains;
* Absence of autonomous drainage system;
* Patient not extubated at the end of the procedure;
* Early reoperation, before drain removal, due to complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The eligible study population will consist of patients aged 18 years and older undergoing major lung resection by conventional or robotic thoracoscopy.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
correlation between intraoperative air leak volume and post-operative air leakage volume | From enrollment to the study completion at 4 weeks
  The primary endpoint is the correlation between intraoperative air leak volume, measured by the ventilator, and postoperative air leak volume, measured by the digitalized autonomous drainage system on the patient's postoperative drain after extubation.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Madalina GRIGOROIU, Principal Investigator — Hôpital Privé d'Antony

IPD SHARING:
Plan to Share IPD: Undecided